CLINICAL TRIAL: NCT02275780
Title: A Phase 3 Multicenter, Double-Blind, Randomized, Active Comparator-Controlled Clinical Trial to Evaluate the Safety and Efficacy of Doravirine (MK-1439) 100 mg Once Daily Versus Darunavir 800 mg Once Daily Plus Ritonavir 100 mg Once Daily, Each in Combination With TRUVADA™ or EPZICOM™/KIVEXA™, in Treatment-Naïve HIV-1 Infected Subjects
Brief Title: Safety and Efficacy of Doravirine (MK-1439) in Participants With Human Immunodeficiency Virus 1 (HIV-1) (MK-1439-018)
Acronym: DRIVE-FORWARD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1439-018; MK-1439-018 (Other: MSD Protocol Number); 2014-001127-69 (EudraCT Number)
Record Dates: First submitted 2014-10-23; First posted 2014-10-27 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: HIV-1
MeSH Terms: interventions — doravirine; Darunavir; Ritonavir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doravirine 100 mg (Experimental): Double-blind Doravirine 100 mg administered orally (p.o.) once daily (q.d.) + investigator selected TRUVADA™ or EPZICOM™/KIVEXA™ administered p.o. q.d. for 96 weeks in the Base Study. Eligible participants may continue in Study Extension 1 with open-label Doravirine 100 mg administered p.o. q.d. + investigator selected TRUVADA™ or EPZICOM™/KIVEXA™ administered p.o., q.d. for an additional 96 weeks. Eligible participants may continue to receive the Doravirine regimen in Study Extension 2 until Doravirine becomes locally available, or for an additional 96 weeks, whichever comes first. Eligible participants may continue to receive the Doravirine regimen in Study Extension 3 until Doravirine becomes locally available, or for an additional 96 weeks, whichever comes first.
  Interventions: Drug: Doravirine; Drug: TRUVADA™ or EPZICOM™/KIVEXA™
- Darunavir 800 mg and Ritonavir 100 mg (Active Comparator): Double-blind Darunavir 800 mg and Ritonavir 100 mg administered p.o. q.d. + investigator selected TRUVADA™ or EPZICOM™/KIVEXA™ administered p.o. q.d. for 96 weeks. Eligible participants may continue in Study Extension 1 with open-label Doravirine 100 mg administered p.o. q.d. + investigator selected TRUVADA™ or EPZICOM™/KIVEXA™ administered p.o. q.d. for an additional 96 weeks. Eligible participants may continue to receive the Doravirine regimen in Study Extension 2 until Doravirine becomes locally available, or for an additional 96 weeks, whichever comes first. Eligible participants may continue to receive the Doravirine regimen in Study Extension 3 until Doravirine becomes locally available, or for an additional 96 weeks, whichever comes first.
  Interventions: Drug: Doravirine; Drug: Darunavir; Drug: Ritonavir; Drug: TRUVADA™ or EPZICOM™/KIVEXA™

INTERVENTIONS:
Drug: Doravirine — Doravirine 100 mg tablet administered p.o. q.d.
Drug: Darunavir — Darunavir 800 mg tablet administered p.o. q.d.
  Arms: Darunavir 800 mg and Ritonavir 100 mg
Drug: Ritonavir — Ritonavir 100 mg tablet administered p.o. q.d.
  Arms: Darunavir 800 mg and Ritonavir 100 mg
Drug: TRUVADA™ or EPZICOM™/KIVEXA™ — The investigator selects either TRUVADA™, a tablet containing 200 mg emtricitabine and 300 mg tenofovir disoproxil fumarate p.o. q.d. or EPZICOM™/KIVEXA™, a tablet containing 600 mg abacavir sulfate and 300 mg lamivudine, p.o. q.d.

SUMMARY:
To establish a new treatment option for treatment-naïve participants with HIV-1, the efficacy and safety of doravirine will be determined relative to a protease inhibitor (PI). Participants will receive double-blind treatment during the 96-week Base Study. Eligible participants in either of the Base Study groups will continue to receive the doravirine-containing regimen open label for an additional 96 weeks in the Study Extension 1. Eligible participants who are deriving benefit will continue in Study Extension 2 to receive the doravirine-containing regimen open label until doravirine becomes locally available or for an additional 96 weeks, whichever comes first. The primary hypothesis is that doravirine 100 mg once a day (q.d.) is non-inferior to darunavir/ritonavir (800 mg/100 mg) q.d., each in combination with TRUVADA™ or EPZICOM™/KIVEXA™, as assessed by the proportion of participants with HIV-1 ribonucleic acid (RNA) <50 copies/mL at Week 48. If non-inferiority is established, then the superiority of doravirine 100 mg q.d. compared to darunavir/ ritonavir (800 mg/100 mg) q.d. will be assessed.

DETAILED DESCRIPTION:
Participants in Australia, Russia, and South Africa who are deriving benefit from MK-1439A are also eligible to continue receiving study drug during Study Extension 3, which will last for 2 years or until drug is available locally, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Is HIV-1 positive and has HIV treatment indicated based on physician assessment.
* Has received no (0 days of) antiretroviral therapy (ART), including investigational antiretroviral agents.
* Is considered clinically stable with no signs or symptoms of active infection for at least 2 weeks prior to the start of treatment.
* Female is highly unlikely to become pregnant, or male is highly unlikely to impregnate a partner because they are not of reproductive potential, or agree to practice abstinence or use acceptable contraception for up to 14 days after the last dose of study drug.
* Eligibility for the Study Extension 1 at the Week 96 visit: 1) completed the Week 96 visit, 2) derived benefit from participation through Week 96 in the opinion of the investigator, 3) is a clinically-appropriate candidate for an additional 96 weeks of treatment with the Study Extension regimen.
* Eligibility for the Study Extension 2 at the Week 192 visit: 1) completed the Week 192 visit, 2) derived benefit from participation through Week 192 in the opinion of the investigator, 3) is a clinically-appropriate candidate for 96 weeks of treatment with the Study Extension regimen.

Exclusion Criteria:

* Uses or has had a recent history of using recreational or illicit drugs.
* Has been treated for a viral infection other than HIV-1, such as hepatitis B, with an agent that is active against HIV-1.
* Has documented or known resistance to study drugs including doravirine, darunavir, ritonavir, emtricitabine, tenofovir, abacavir and/or lamivudine.
* Has participated in a study with an investigational compound/device within the prior month, or anticipates doing so during this study.
* Has used systemic immunosuppressive therapy or immune modulators within the prior 30 days, or anticipates doing so during this study.
* Has significant hypersensitivity or other contraindication to any of the components of the study drugs.
* Has a current (active) diagnosis of acute hepatitis due to any cause.
* Is pregnant, breastfeeding or expecting to conceive at any time during the study.
* Female who expects to donate eggs, or male who expects to donate sperm at any time during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 769 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2016-09-29 (Actual); Study Completion 2023-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Orkin C, Koethe JR, Kumar PN, Sklar P, Xu ZJ, Plank RM, Greaves W, Lahoulou R. Factors Associated With Weight Change After Continuing or Switching to a Doravirine-based Regimen. Open Forum Infect Dis. 2025 Nov 20;12(11):ofaf639. doi: 10.1093/ofid/ofaf639. eCollection 2025 Nov. PMID 41280318
- [Derived] Hsue PY, Behrens GMN, Xu ZJ, Zhao Y, Cmar J, Lahoulou R, Campo RE, Plank RM. Cardiovascular Risk Assessment Using the Atherosclerotic Cardiovascular Disease Risk Score Model after Continuing or Switching to a Doravirine-Based HIV Treatment Regimen. J Acquir Immune Defic Syndr. 2026 Feb 1;101(2):208-213. doi: 10.1097/QAI.0000000000003778. PMID 41081774
- [Derived] Walmsley SL, Kumar PN, Orkin C, Thompson M, Squires K, Xu ZJ, Greaves W, Plank RM, Whiteside Y, Lahoulou R. Efficacy and Safety of Doravirine-based Regimens by Sex and Race: Long-term Results From Three Phase 3 Clinical Trials. Open Forum Infect Dis. 2025 Jul 16;12(7):ofaf356. doi: 10.1093/ofid/ofaf356. eCollection 2025 Jul. PMID 40672760
- [Derived] Moyle G, Meng F, Wan H, Sklar P, Plank RM, Lahoulou R. Brief Report: Resolution of Neuropsychiatric Adverse Events After Switching to a Doravirine-Based Regimen in the Open-Label Extensions of the DRIVE-AHEAD and DRIVE-FORWARD Trials. J Acquir Immune Defic Syndr. 2025 May 1;99(1):81-86. doi: 10.1097/QAI.0000000000003599. PMID 39748155
- [Derived] Orkin C, Molina JM, Cahn P, Lombaard J, Supparatpinyo K, Kumar S, Campbell H, Wan H, Teal V, Jin Xu Z, Asante-Appiah E, Sklar P, Teppler H, Lahoulou R; DRIVE-FORWARD and DRIVE-AHEAD collaborators. Safety and efficacy of doravirine as first-line therapy in adults with HIV-1: week 192 results from the open-label extensions of the DRIVE-FORWARD and DRIVE-AHEAD phase 3 trials. Lancet HIV. 2024 Feb;11(2):e75-e85. doi: 10.1016/S2352-3018(23)00258-8. Epub 2023 Dec 20. PMID 38141637
- [Derived] Molina JM, Squires K, Sax PE, Cahn P, Lombaard J, DeJesus E, Lai MT, Rodgers A, Lupinacci L, Kumar S, Sklar P, Hanna GJ, Hwang C, Martin EA; DRIVE-FORWARD trial group. Doravirine versus ritonavir-boosted darunavir in antiretroviral-naive adults with HIV-1 (DRIVE-FORWARD): 96-week results of a randomised, double-blind, non-inferiority, phase 3 trial. Lancet HIV. 2020 Jan;7(1):e16-e26. doi: 10.1016/S2352-3018(19)30336-4. Epub 2019 Nov 15. PMID 31740348
- [Derived] Orkin C, Molina JM, Lombaard J, DeJesus E, Rodgers A, Kumar S, Martin E, Hanna G, Hwang C. Once-daily Doravirine in Human Immunodeficiency Virus Type 1-Infected, Antiretroviral-naive Adults: An Integrated Efficacy Analysis. Clin Infect Dis. 2020 Mar 17;70(7):1344-1352. doi: 10.1093/cid/ciz424. PMID 31121015
- [Derived] Thompson M, Orkin C, Molina JM, Sax P, Cahn P, Squires K, Xu X, Rodgers A, Kumar S, Teppler H, Martin E, Hanna G, Hwang C. Once-daily Doravirine for Initial Treatment of Adults Living With Human Immunodeficiency Virus-1: An Integrated Safety Analysis. Clin Infect Dis. 2020 Mar 17;70(7):1336-1343. doi: 10.1093/cid/ciz423. PMID 31121013
- [Derived] Molina JM, Squires K, Sax PE, Cahn P, Lombaard J, DeJesus E, Lai MT, Xu X, Rodgers A, Lupinacci L, Kumar S, Sklar P, Nguyen BY, Hanna GJ, Hwang C; DRIVE-FORWARD Study Group. Doravirine versus ritonavir-boosted darunavir in antiretroviral-naive adults with HIV-1 (DRIVE-FORWARD): 48-week results of a randomised, double-blind, phase 3, non-inferiority trial. Lancet HIV. 2018 May;5(5):e211-e220. doi: 10.1016/S2352-3018(18)30021-3. Epub 2018 Mar 25. PMID 29592840
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26091&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1027 participants were screened and 769 were randomized.
Groups:
- Doravirine 100 mg: Double-blind Doravirine 100 mg administered orally (p.o.) once daily (q.d.) + investigator-selected TRUVADA™ or EPZICOM™/KIVEXA™ administered p.o. q.d. for 96 weeks in the Base Study. Eligible participants continued in Study Extension 1 with open-label Doravirine 100 mg administered p.o. q.d. + investigator-selected TRUVADA™ or EPZICOM™/ KIVEXA™ administered p.o. q.d. for an additional 96 weeks. Eligible participants continued to receive the Doravirine regimen in Study Extension 2 for an additional 96 weeks, and in Study Extension 3 for an additional 96 weeks.
- Daurunavir 800 mg + Ritonavir 100 mg → Doravirine 100 mg: Double-blind Darunavir 800 mg and Ritonavir 100 mg administered p.o. q.d. + investigator-selected TRUVADA™ or EPZICOM™/ KIVEXA™ administered p.o. q.d. for 96 weeks in the Base Study. Eligible participants continued in Study Extension 1 with open-label Doravirine 100 mg administered p.o. q.d. + investigator-selected TRUVADA™ or EPZICOM™/ KIVEXA™ administered p.o. q.d. for an additional 96 weeks. Eligible participants continued to receive the Doravirine regimen in Study Extension 2 for an additional 96 weeks, and in Study Extension 3 for an additional 96 weeks.
Period: Base Study: 96 Weeks
Arm/Group | Doravirine 100 mg | Daurunavir 800 mg + Ritonavir 100 mg → Doravirine 100 mg
Started | 385 | 384
Treated | 383 | 383
Completed | 292 | 273
Not Completed | 93 | 111
Not completed — Adverse Event | 6 | 14
Not completed — Death | 3 | 1
Not completed — Lack of Efficacy | 21 | 32
Not completed — Lost to Follow-up | 28 | 24
Not completed — Protocol Violation | 1 | 6
Not completed — Withdrawal by Subject | 19 | 22
Not completed — Noncompliance with drug | 9 | 6
Not completed — Physician Decision | 2 | 4
Not completed — Pregnancy | 2 | 1
Not completed — Randomized not treated | 2 | 1
Period: Study Extension 1: Week 96 to Week 192
Arm/Group | Doravirine 100 mg | Daurunavir 800 mg + Ritonavir 100 mg → Doravirine 100 mg
Started | 259 (Study Extension 1 was optional; not all eligible participants enrolled.) | 233 (Study Extension was optional; not all eligible participants enrolled.)
Completed | 210 | 190
Not Completed | 49 | 43
Not completed — Adverse Event | 6 | 1
Not completed — Availability of study medication locally | 2 | 0
Not completed — Lack of Efficacy | 8 | 11
Not completed — Lost to Follow-up | 8 | 7
Not completed — Non-compliance with study drug | 1 | 2
Not completed — Physician Decision | 3 | 7
Not completed — Pregnancy | 2 | 1
Not completed — Withdrawal by Subject | 19 | 14
Period: Study Extension 2: Week 192 to Week 288
Arm/Group | Doravirine 100 mg | Daurunavir 800 mg + Ritonavir 100 mg → Doravirine 100 mg
Started | 148 (Study Extension 2 was optional; not all eligible participants enrolled.) | 129 (Study Extension 2 was optional; not all eligible participants enrolled.)
Completed | 101 | 91
Not Completed | 47 | 38
Not completed — Adverse Event | 0 | 1
Not completed — Availability of study medication locally | 38 | 29
Not completed — Lack of Efficacy | 2 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Non-compliance with study drug | 2 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 4 | 3
Period: Study Extension 3: Week 288 to Week 384
Arm/Group | Doravirine 100 mg | Daurunavir 800 mg + Ritonavir 100 mg → Doravirine 100 mg
Started | 50 (Study Extension 3 was optional; not all eligible participants enrolled.) | 36 (Study Extension 3 was optional; not all eligible participants enrolled.)
Completed | 36 | 23
Not Completed | 14 | 13
Not completed — Availability of study medication locally | 6 | 6
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 3
Not completed — Non-compliance with study drug | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Doravirine 100 mg: Double-blind Doravirine 100 mg administered p.o. q.d. + investigator-selected TRUVADA™ or EPZICOM™/KIVEXA™ administered p.o. q.d. for 96 weeks in the Base Study.
- Daurunavir 800 mg + Ritonavir 100 mg: Double-blind Darunavir 800 mg and Ritonavir 100 mg administered p.o. q.d. + investigator-selected TRUVADA™ or EPZICOM™/ KIVEXA™ administered p.o. q.d. for 96 weeks in the Base Study.
- Total: Total of all reporting groups
Arm/Group | Doravirine 100 mg | Daurunavir 800 mg + Ritonavir 100 mg | Total
Number analyzed (Participants) | 385 | 384 | 769
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.9 (10.7) | 35.7 (10.7) | 35.3 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 58 | 123
  Male | 320 | 326 | 646
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 93 | 86 | 179
  Not Hispanic or Latino | 286 | 291 | 577
  Unknown or Not Reported | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 7 | 7 | 14
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 87 | 89 | 176
  White | 281 | 280 | 561
  More than one race | 6 | 2 | 8
  Unknown or Not Reported | 0 | 1 | 1
Mean Cluster of Differentiation 4 (CD4+) T-cell Count [Mean (Standard Deviation); unit: Cells/mm^3] — CD4+ T-cell count was quantified by a central laboratory using a commercially available assay. Population: Participants with baseline data
  Cells/mm^3
    number analyzed (Participants) | 383 | 383 | 766
    (all) | 432.6 (208.4) | 411.9 (229.6) | 422.2 (219.4)
Plasma HIV-1 RNA [Median (Full Range); unit: Copies/mL] — Plasma HIV-1 RNA levels were quantified with the Abbott RealTime HIV-1 Assay. Population: Participants with baseline data
  Copies/mL
    number analyzed (Participants) | 383 | 382 | 765
    (all) | 27073.0 [105 to 2776658] | 27357.0 [235 to 3272236] | 27073.0 [105 to 3272236]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Plasma HIV-1 RNA <50 Copies/mL at Week 48
Description: The percentage of participants in each arm achieving HIV-1 RNA levels <50 copies/mL at Week 48 was determined. Plasma HIV-1 RNA levels were quantified with the Abbott RealTime HIV-1 Assay. Data were handled according to the US Food and Drug Administration (FDA) "snapshot" approach and all missing data were considered treatment failures, regardless of the reason.
Time Frame: Week 48
Population: All randomized participants who received at least 1 dose of study drug
Measure: Number; unit: Percentage of participants
Arm/Group | Doravirine 100 mg | Daurunavir 800 mg + Ritonavir 100 mg
Number analyzed (Participants) | 383 | 383
Percentage of participants | 83.8 | 79.9
Statistical Analysis 1: Comparison: Doravirine 100 mg vs Daurunavir 800 mg + Ritonavir 100 mg; Test type: Non-Inferiority — Doravirine is concluded to be non-inferior to darunavir + ritonavir if the lower bound of the 95% CI for the difference in percent response is above -10 percentage points; Treatment Difference = 3.913, 95% CI 2-sided [-1.590 to 9.415] — Stratum-adjusted Mantel-Haenszel method with the difference weighted by the harmonic mean of sample size per arm for each stratum

2. Secondary Outcome: Percentage of Participants Achieving Plasma HIV-1 RNA <50 Copies/mL at Week 96
Description: The percentage of participants in each arm achieving HIV-1 RNA levels <50 copies/mL at Week 96 was determined. Plasma HIV-1 RNA levels were quantified with the Abbott RealTime HIV-1 Assay. Data were handled according to the US Food and Drug Administration (FDA) "snapshot" approach and all missing data were considered treatment failures, regardless of the reason.
Time Frame: Week 96
Population: All randomized participants who received at least 1 dose of study drug and had data for the outcome measure. Participants with missing HIV-1 RNA due to an Abbott RealTime manufacturing agent recall were excluded from the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Doravirine 100 mg | Daurunavir 800 mg + Ritonavir 100 mg
Number analyzed (Participants) | 379 | 376
Percentage of participants | 73.1 | 66.0
Statistical Analysis 1: Comparison: Doravirine 100 mg vs Daurunavir 800 mg + Ritonavir 100 mg; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Treatment Difference = 7.082, 95% CI 2-sided [0.508 to 13.656] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in Mean CD4+ T-cell Count at Week 48
Description: CD4+ T-cell counts were quantified by a central laboratory using a commercially available assay.
Time Frame: Baseline and Week 48
Population: All randomized participants who received at least 1 dose of study drug and had data for the outcome measure. Baseline values were carried forward for participants who discontinued therapy due to lack of efficacy.
Measure: Mean (95% Confidence Interval); unit: Cells/mm^3
Arm/Group | Doravirine 100 mg | Daurunavir 800 mg + Ritonavir 100 mg
Number analyzed (Participants) | 363 | 353
Cells/mm^3 | 192.7 [171.5 to 213.9] | 185.6 [167.5 to 203.6]
Statistical Analysis 1: Comparison: Doravirine 100 mg vs Daurunavir 800 mg + Ritonavir 100 mg; Test type: Other; Mean treatment difference = 7.1, 95% CI 2-sided [-20.8 to 35.0] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline in Mean CD4+ T-cell Count at Week 96
Description: CD4+ T-cell counts were quantified by a central laboratory using a commercially available assay.
Time Frame: Baseline and Week 96
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Cells/mm^3
Arm/Group | Doravirine 100 mg | Daurunavir 800 mg + Ritonavir 100 mg
Number analyzed (Participants) | 342 | 327
Cells/mm^3 | 224.1 [200.8 to 247.4] | 206.7 [184.9 to 228.5]
Statistical Analysis 1: Comparison: Doravirine 100 mg vs Daurunavir 800 mg + Ritonavir 100 mg; Test type: Other; Mean treatment difference = 17.4, 95% CI 2-sided [-14.5 to 49.3] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Mean Change From Baseline in Fasting Low Density Lipoprotein Cholesterol (LDL-C) at Week 48
Description: Serum LDL-C was determined after an overnight fast. Change from Baseline was analyzed using ANCOVA models with terms for Baseline lipid level and treatment group. The Last Observation Carry Forward (LOCF) approach was applied for missing data or data collected after modifying lipid-lowering therapy.
Time Frame: Baseline and Week 48
Population: All randomized participants who received at least 1 dose of study drug and had a measurement at Baseline and at the time point assessed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Doravirine 100 mg | Daurunavir 800 mg + Ritonavir 100 mg
Number analyzed (Participants) | 326 | 318
mg/dL
  Baseline | 91.10 (28.61) | 91.76 (30.36)
  Change from Baseline | -4.51 (20.64) | 9.92 (27.31)
Statistical Analysis 1: Comparison: Doravirine 100 mg vs Daurunavir 800 mg + Ritonavir 100 mg; Test type: Other; p < 0.0001, ANCOVA; Terms for Baseline lipid level and treatment group; Treatment Difference (mg/dL) = -14.61, 95% CI 2-sided [-18.15 to -11.06]

6. Secondary Outcome: Mean Change From Baseline in Fasting Non-High Density Lipoprotein Cholesterol (Non-HDL-C) at Week 48
Description: Serum non-HDL-C was determined after an overnight fast. Change from Baseline was analyzed using ANCOVA models with terms for Baseline lipid level and treatment group. The LOCF approach was applied for missing data or data collected after modifying lipid-lowering therapy.
Time Frame: Baseline and Week 48
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Doravirine 100 mg | Daurunavir 800 mg + Ritonavir 100 mg
Number analyzed (Participants) | 329 | 325
mg/dL
  Baseline | 113.34 (34.25) | 114.44 (35.01)
  Change from Baseline | -5.30 (23.28) | 13.75 (31.08)
Statistical Analysis 1: Comparison: Doravirine 100 mg vs Daurunavir 800 mg + Ritonavir 100 mg; Test type: Other; p < 0.0001, ANCOVA; Terms for Baseline lipid level and treatment group; Treatment Difference (mg/dL) = -19.34, 95% CI 2-sided [-23.33 to -15.35]

7. Secondary Outcome: Mean Change From Baseline in Fasting High Density Lipoprotein Cholesterol (HDL-C) at Week 48
Description: Serum HDL-C was determined after an overnight fast. Change from Baseline was analyzed using ANCOVA models with terms for Baseline lipid level and treatment group. The LOCF approach was applied for missing data or data collected after modifying lipid-lowering therapy.
Time Frame: Baseline and Week 48
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Doravirine 100 mg | Daurunavir 800 mg + Ritonavir 100 mg
Number analyzed (Participants) | 329 | 325
mg/dL
  Baseline | 43.58 (12.99) | 43.27 (13.96)
  Change from Baseline | 3.94 (10.66) | 4.15 (11.01)

8. Secondary Outcome: Mean Change From Baseline in Fasting Total Cholesterol at Week 48
Description: Serum total cholesterol was determined after an overnight fast. Change from Baseline was analyzed using ANCOVA models with terms for Baseline lipid level and treatment group. The LOCF approach was applied for missing data or data collected after modifying lipid-lowering therapy.
Time Frame: Baseline and Week 48
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Daurunavir 800 mg + Ritonavir 100 mg → Doravirine 100 mg: Double-blind Darunavir 800 mg and Ritonavir 100 mg administered p.o. q.d. + investigator-selected TRUVADA™ or EPZICOM™/ KIVEXA™ administered p.o. q.d. for 96 weeks in the Base Study.
Arm/Group | Doravirine 100 mg | Daurunavir 800 mg + Ritonavir 100 mg → Doravirine 100 mg
Number analyzed (Participants) | 329 | 325
mg/dL
  Baseline | 156.92 (35.82) | 157.71 (37.34)
  Change from Baseline | -1.37 (25.47) | 17.90 (33.95)

9. Secondary Outcome: Mean Change From Baseline in Fasting Triglyceride at Week 48
Description: Serum triglyceride was determined after an overnight fast. Change from Baseline was analyzed using ANCOVA models with terms for Baseline lipid level and treatment group. The LOCF approach was applied for missing data or data collected after modifying lipid-lowering therapy.
Time Frame: Baseline and Week 48
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Doravirine 100 mg | Daurunavir 800 mg + Ritonavir 100 mg
Number analyzed (Participants) | 329 | 325
mg/dL
  Baseline | 111.16 (75.31) | 117.02 (97.30)
  Change from Baseline | -3.14 (68.81) | 21.97 (92.59)

10. Secondary Outcome: Percentage of Participants With Any Adverse Event
Description: An adverse event (AE) is defined as any untoward medical occurrence in a study participant and which does not necessarily have to have a causal relationship to treatment. An adverse event can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the study treatment or protocol-specified procedure, whether or not considered related to study treatment or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the study treatment is also an AE. The percentage of participants with any AE was assessed.
Time Frame: Up to 98 weeks
Population: All randomized participants who received at least 1 dose of study drug
Measure: Number; unit: Percentage of participants
Arm/Group | Doravirine 100 mg | Daurunavir 800 mg + Ritonavir 100 mg
Number analyzed (Participants) | 383 | 383
Percentage of participants | 84.6 | 82.8

11. Secondary Outcome: Percentage of Participants With Any Serious Adverse Event
Description: A serious adverse event is an AE that results in death, is life threatening, results in persistent or significant disability or incapacity, results in or prolongs a hospitalization, is a congenital anomaly or birth defect, is a cancer, is associated with an overdose, or is another important medical event. The percentage of participants with any SAE was assessed.
Time Frame: Up to 98 weeks
Population: All randomized participants who received at least 1 dose of study drug
Measure: Number; unit: Percentage of participants
Arm/Group | Doravirine 100 mg | Daurunavir 800 mg + Ritonavir 100 mg
Number analyzed (Participants) | 383 | 383
Percentage of participants | 7.0 | 8.6

12. Secondary Outcome: Percentage of Participants With Any Drug-related Adverse Event
Description: The investigator was to determine if an AE had a reasonable possibility of a relationship to the study drug. The percentage of participants with any drug-related AE was assessed.
Time Frame: Up to 98 weeks
Population: All randomized participants who received at least 1 dose of study drug
Measure: Number; unit: Percentage of participants
Arm/Group | Doravirine 100 mg | Daurunavir 800 mg + Ritonavir 100 mg
Number analyzed (Participants) | 383 | 383
Percentage of participants | 32.1 | 32.1

13. Secondary Outcome: Percentage of Participants With Any Drug-related Serious Adverse Event
Description: The percentage of participants with any drug-related SAE was assessed.
Time Frame: Up to 98 weeks
Population: All randomized participants who received at least 1 dose of study drug
Measure: Number; unit: Percentage of participants
Arm/Group | Doravirine 100 mg | Daurunavir 800 mg + Ritonavir 100 mg
Number analyzed (Participants) | 383 | 383
Percentage of participants | 0.3 | 0.3

14. Secondary Outcome: Percentage of Participants Who Discontinued Study Treatment Due to an Adverse Event
Description: The percentage of participants who discontinued study treatment due to an AE was assessed.
Time Frame: Up to 96 weeks
Population: All randomized participants who received at least 1 dose of study drug
Measure: Number; unit: Percentage of participants
Arm/Group | Doravirine 100 mg | Daurunavir 800 mg + Ritonavir 100 mg
Number analyzed (Participants) | 383 | 383
Percentage of participants | 1.6 | 3.4

15. Secondary Outcome: Percentage of Participants Achieving Plasma HIV-1 RNA <40 Copies/mL at Week 48
Description: The percentage of participants in each arm achieving HIV-1 RNA levels <40 copies/mL at Week 48 was determined. Plasma HIV-1 RNA levels were quantified with the Abbott RealTime HIV-1 Assay. Data were handled according to the US Food and Drug Administration (FDA) "snapshot" approach and all missing data were considered treatment failures, regardless of the reason.
Time Frame: Week 48
Population: All randomized participants who received at least 1 dose of study drug
Measure: Number; unit: Percentage of participants
Arm/Group | Doravirine 100 mg | Daurunavir 800 mg + Ritonavir 100 mg
Number analyzed (Participants) | 383 | 383
Percentage of participants | 83.3 | 79.1
Statistical Analysis 1: Comparison: Doravirine 100 mg vs Daurunavir 800 mg + Ritonavir 100 mg; Test type: Other; Treatment Difference = 4.169, 95% CI 2-sided [-1.404 to 9.743] — [estimate comment as in outcome 1, analysis 1]

16. Secondary Outcome: Percentage of Participants Achieving Plasma HIV-1 RNA <40 Copies/mL at Week 96
Description: The percentage of participants in each arm achieving HIV-1 RNA levels <40 copies/mL at Week 96 was determined. Plasma HIV-1 RNA levels were quantified with the Abbott RealTime HIV-1 Assay. Data were handled according to the US Food and Drug Administration (FDA) "snapshot" approach and all missing data were considered treatment failures, regardless of the reason.
Time Frame: Week 96
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Doravirine 100 mg | Daurunavir 800 mg + Ritonavir 100 mg
Number analyzed (Participants) | 379 | 376
Percentage of participants | 72.0 | 64.4
Statistical Analysis 1: Comparison: Doravirine 100 mg vs Daurunavir 800 mg + Ritonavir 100 mg; Test type: Other; Treatment Difference = 7.606, 95% CI 2-sided [0.980 to 14.232] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to Week 386
Description: The analysis population for All-Cause Mortality included all randomized participants. The analysis population for Serious and Other Adverse Events included all participants who received at least 1 dose of study drug.
Groups:
- Doravirine 100 mg: Double-blind Doravirine 100 mg administered p.o. q.d. + investigator-selected TRUVADA™ or EPZICOM™/KIVEXA™ administered p.o. q.d. for 96 weeks in the Base Study. Eligible participants continued in Study Extension 1 with open-label Doravirine 100 mg administered p.o. q.d. + investigator-selected TRUVADA™ or EPZICOM™/ KIVEXA™ administered p.o. q.d. for an additional 96 weeks. Eligible participants continued to receive the Doravirine regimen in Study Extension 2 for an additional 96 weeks, and in Study Extension 3 for an additional 96 weeks.
Arm/Group | Doravirine 100 mg | Daurunavir 800 mg + Ritonavir 100 mg → Doravirine 100 mg
All-Cause Mortality (participants affected / at risk) | 3/385 | 3/384
Serious Adverse Events (participants affected / at risk) | 45/383 | 49/383
Other Adverse Events (participants affected / at risk) | 264/383 | 247/383
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doravirine 100 mg (N=383) | Daurunavir 800 mg + Ritonavir 100 mg → Doravirine 100 mg (N=383)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal skin tags (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis necrotising (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (5)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Acute hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (3) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Chronic hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Fournier's gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis shigella (Infections and infestations) | 0 (0) | 1 (1)
Herpes oesophagitis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Keratouveitis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis tuberculous (Infections and infestations) | 0 (0) | 1 (1)
Neurosyphilis (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pilonidal disease (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 2 (2)
Rectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Scrotal abscess (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 2 (2)
Tuberculosis of central nervous system (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Rectal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Bell's palsy (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Osmotic demyelination syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Post abortion haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Drug dependence (Psychiatric disorders) | 1 (2) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Schizoaffective disorder depressive type (Psychiatric disorders) | 0 (0) | 1 (1)
Substance-induced mood disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug abuser (Social circumstances) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Femoral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doravirine 100 mg (N=383) | Daurunavir 800 mg + Ritonavir 100 mg → Doravirine 100 mg (N=383)
Abdominal pain (Gastrointestinal disorders) | 20 (22) | 20 (25)
Abdominal pain upper (Gastrointestinal disorders) | 27 (30) | 15 (18)
Diarrhoea (Gastrointestinal disorders) | 72 (87) | 100 (136)
Nausea (Gastrointestinal disorders) | 52 (65) | 54 (64)
Vomiting (Gastrointestinal disorders) | 20 (32) | 12 (14)
Fatigue (General disorders) | 38 (40) | 28 (30)
Pyrexia (General disorders) | 21 (21) | 10 (10)
Bronchitis (Infections and infestations) | 31 (43) | 37 (42)
Gastroenteritis (Infections and infestations) | 22 (25) | 23 (28)
Influenza (Infections and infestations) | 24 (29) | 16 (20)
Nasopharyngitis (Infections and infestations) | 61 (110) | 61 (102)
Syphilis (Infections and infestations) | 29 (39) | 39 (47)
Upper respiratory tract infection (Infections and infestations) | 64 (115) | 40 (59)
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 (29) | 22 (27)
Back pain (Musculoskeletal and connective tissue disorders) | 37 (45) | 13 (16)
Dizziness (Nervous system disorders) | 25 (28) | 24 (28)
Headache (Nervous system disorders) | 63 (106) | 59 (92)
Insomnia (Psychiatric disorders) | 27 (27) | 23 (27)
Cough (Respiratory, thoracic and mediastinal disorders) | 38 (48) | 14 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-23): https://cdn.clinicaltrials.gov/large-docs/80/NCT02275780/Prot_SAP_000.pdf